CLINICAL TRIAL: NCT03981497
Title: Retrospective and Perspective Analysis of Short, Medium and Long Term Clinical Performance of Patients Undergoing MicrowaveThermal Ablation for Treatment of Small Renal Tumors and Primary and Secondary Liver Neoplasms
Brief Title: Microwave Ablation for Treatment of Small Renal Tumors and Primary and Secondary Liver Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Francesco De Cobelli (Other)
Responsible Party: Sponsor-Investigator, Francesco De Cobelli, Professor of Radiology, Clinical and Experimental Radiology, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: MWA-01
Record Dates: First submitted 2019-05-27; First posted 2019-06-10 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Liver Cancer; Liver Metastasis Colon Cancer; Kidney Cancer; Renal Cell Carcinoma
Keywords: MWA
MeSH Terms: conditions — Liver Neoplasms; Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Small Renal Tumors: Subjects with small renal tumors (SRT) ad described by current ESMO (European Society for Medical Oncology) guidelines who are candidates for MWA
  Interventions: Procedure: Microwave ablation (MWA)
- Primary and Secondary Liver cancer: Primary liver tumors: subjects who are candidates for MWA with nodules ≤ 3 cm Liver metastases: subjects who are candidates for MWA with nodules less than ≤ 3 cm
  Interventions: Procedure: Microwave ablation (MWA)

INTERVENTIONS:
Procedure: Microwave ablation (MWA) — Thermal ablation

SUMMARY:
The goal of this observational study is to collect data on efficacy and safety of microwave ablation (MWA) used to treat subjects with primary and secondary liver malignancies and renal malignancies. The main question it aims to evaluate the short, medium and long-term clinical course of patients treated with MWA.

Participants will not alter their normal clinical and therapeutic practice, due to the observational nature of the study, and all data regarding microwave treatments will be collected (including demographic data). follow their normal clinical and therapeutic path

DETAILED DESCRIPTION:
Observational, retrospective and prospective, monocentric study. The objective is to evaluate the short, medium and long-term clinical course of patients undergoing microwave ablation (MWA) for small renal tumors and primary and secondary liver neoplasms. Evaluation of clinical efficacy (progression free survival),safety and technical outcome of microwave ablation as well as clinical outcome of the procedure will be evaluated.At the end of the follow-up periods, the data collected will be compared with those available in the literature on MWA, cryoablation (CA), radiofrequency ablation (RFA) and surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years with primary or secondary liver tumors or small kidney tumors that are not candidates for surgery or cannot be radically resected by surgery alone
* Primary liver cancer: up to three liver nodules ≤ 3 cm
* Secondary hepatic tumours: up to nodules ≤ 3 cm provided that the objective is complete hepatic clearance Renal tumours: single or multiple (von Hippel Lindau syndrome), < 4 cm

Exclusion Criteria:

* pregnant women
* non-manageable coagulopathies
* Extended extrahepatic or extrarenal disease
* for liver ablation: presence of bilio-digestive anastomosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with indication of laparoscopic or percutaneous ablation of primary or secondary liver tumors and small primary kidney tumors (according to ESMO guidelines).
  All patients will follow their normal therapeutic procedure and no examination will be added to what is already provided for in the normal management of patients suffering from these diseases.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Tumor Progression Free Survival | From date of ablation until death from any cause; evaluated up to 5 years
  Based on imaging evidence of tumor reccurence at site of ablation (within 5mm of ablation margins)
Time to Local Progression | From date of ablation until death from any cause; evaluated up to 5 years
  Time from ablation to imaging evidence of tumor reccurence at site of ablation (within 5mm of ablation margins)

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of ablation until death from any cause; evaluated up to 5 years
  From date of ablation until death for any cause
Progression Free Survival (PFS) | From date of ablation until death from any cause; evaluated up to 5 years
  From date of ablation until any documented evidence of tumor progression at any site
Organ specific Progression Free Survival (PFS) | From date of ablation until death from any cause; evaluated up to 5 years
  From date of ablation until any documented evidence of tumor progression at the ablated organ (including reccurence at ablation site)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Cobelli F, Marra P, Ratti F, Ambrosi A, Colombo M, Damascelli A, Sallemi C, Gusmini S, Salvioni M, Diana P, Cipriani F, Venturini M, Aldrighetti L, Del Maschio A. Microwave ablation of liver malignancies: comparison of effects and early outcomes of percutaneous and intraoperative approaches with different liver conditions : New advances in interventional oncology: state of the art. Med Oncol. 2017 Apr;34(4):49. doi: 10.1007/s12032-017-0903-8. Epub 2017 Feb 20. PMID 28220346
- [Derived] di Gaeta E, Olivieri M, Savi A, Magnani P, Canevari C, Gusmini S, Palumbo D, Guazzarotti G, Augello L, Calabrese F, Steidler S, Cipriani F, Rimini M, Casadei-Gardini A, Aldrighetti L, Chiti A, De Cobelli F. Radioembolization for Hepatocellular Carcinoma: a Comparison on Dual-phase Cone-beam CT, Contrast-enhanced CT (CECT) and 99mTc-macroaggregated albumin-SPECT/CT in predicting final distribution volumes and dosimetry of the post-embolization 90Y PET/CT. Radiol Med. 2025 Apr;130(4):474-485. doi: 10.1007/s11547-024-01946-0. Epub 2024 Dec 20. PMID 39707126